CLINICAL TRIAL: NCT07144280
Title: A RANDOMIZED, PHASE 3, OPEN-LABEL STUDY TO EVALUATE PF-08046054/SGN-PDLlV VERSUS DOCETAXEL IN ADULT PARTICIPANTS WITH PREVIOUSLY-TREATED PROGRAMMED CELL DEATH LIGAND 1 (PD-Ll) POSITIVE NON-SMALL-CELL LUNG CANCER (NSCLC)
Brief Title: A Study to Learn About the Study Medicine Called PF-08046054/SGN-PDL1V Versus Docetaxel in Adult Participants With Previously-treated Programmed Cell Death Ligand 1 (PD-L1) Positive Non-Small-Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C5851005; 2025-521281-97-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Carcinoma; Non-Small Cell Lung Cancer Metastatic; Non-Small Cell Lung Carcinoma
Keywords: Non-small cell lung cancer NSCLC; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PF-08046054 monotherapy (Experimental): PF-08046054 monotherapy
  Interventions: Drug: PF-08046054
- Docetaxel monotherapy (Active Comparator): Docetaxel monotherapy
  Interventions: Drug: Docetaxel monotherapy

INTERVENTIONS:
Drug: PF-08046054 — Antibody Drug Conjugate
  Participants will receive PF-08046054, administered as an IV infusion.
  Other Names: SGN-PDL1V
  Arms: PF-08046054 monotherapy
Drug: Docetaxel monotherapy — Participants will receive Docetaxel, administered as an IV infusion.
  Arms: Docetaxel monotherapy

SUMMARY:
The purpose of this study is to understand if PF-08046054 alone works well compared to standard-of-care docetaxel alone in participants with non-small cell lung cancer (NSCLC) with PD-L1 expression greater than or equal to 1% and had cancer progression during or after treatment with PD-L1 or PD-1 inhibitors, platinum-based chemotherapy, and targeted treatment regimen(s) for participants with known actionable genomic alterations (AGAs). Participants in this study must have cancer that has spread through their body or can't be removed with surgery or treated with definitive radiation.

Participants will randomly (like a flip of the coin) be assigned to either the PF-08046054 treatment group or the docetaxel treatment group. Participants in the PF-08046054 treatment group will receive an IV infusion (injected directly into the veins) twice during each 21-day cycle. Participants in the docetaxel treatment group will receive an IV infusion once during each 21-day cycle. Study participation may be up to 5 years if the participant's NSCLC is responding to treatment. The study team will see how each participant is doing with the study treatment during regular visits at the clinic.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed diagnosis of locally advanced, unresectable Stage IIIB and IIIC not eligible for definitive chemoradiotherapy or metastatic (Stage IV: M1a, M1b, or M1c) NSCLC per the American Joint Committee on Cancer (AJCC) Staging Manual, Version 8.0, and the Union for International Cancer Control (UICC) Staging System. Note: Participants with a neuroendocrine component or histology are not eligible.
2. PD-L1 expression on ≥1% of tumor cells based on local immunohistochemistry (IHC) testing with an assay utilizing the anti-PD-L1 monoclonal antibody clones 22C3 or SP263.
3. Participants who have NSCLC with known AGAs are permitted (eg, estimated glomerular filtration rate (EGFR) mutations, anaplastic lymphoma kinase (ALK) translocations).
4. Able to provide any of the following tumor tissues for biomarker analysis:

   * Archival specimen (preferably collected within 12 months after the last anticancer therapy) (see laboratory manual for details); or
   * Fresh tissue from a tumor lesion, if medically feasible.
5. Participants must have received the following therapies and progressed during or relapsed after receiving their most recent prior therapy:

Participants with no known AGAs must fulfill 1 of the following conditions:

* Received a platinum-based combination therapy for the treatment of metastatic or recurrent disease and a PD-L1 or PD-1 monoclonal antibody (concurrently or sequentially with platinum-based chemotherapy), unless contraindicated.
* Experienced disease progression within 6 months of the last dose of platinum-based chemotherapy in the adjuvant, neoadjuvant, or chemoradiotherapy setting and received a PD-L1 or PD-1 monoclonal antibody at any time during the course of treatment.

Participants with known AGAs (eg, EGFR mutations, ALK translocations, or other relevant actionable mutations) must fulfill the following conditions:

* Must have received at least 1 approved AGA-targeted therapy and, in the opinion of the investigator, additional AGA-targeted therapy is not in the best interest of the participant
* Received a platinum-based combination therapy for the treatment of metastatic or recurrent disease, or experienced disease progression within 6 months of the last dose of platinum-based chemotherapy in the adjuvant, neoadjuvant, or chemoradiotherapy setting.
* May have received PD-1 or PD-L1 monoclonal antibody (concurrently or sequentially with platinum-based chemotherapy).

Exclusion Criteria

1. History of another malignancy within 3 years before the first dose of PF-08046054, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death (eg, 5-year overall survival (OS) ≥90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
2. Active central nervous system (CNS) lesions are excluded. Active is defined as untreated or symptomatic requiring corticosteroids >10 mg/day of prednisone equivalent within the previous 14 days.

   Participants with clinically inactive, definitively treated brain metastases (surgery and/or radiotherapy) are eligible if they meet the following criteria:
   * The participant is on a stable dose of ≤10 mg/day of prednisone or equivalent for at least >14 days (if requiring steroid treatment).
   * No evidence of clinical and radiographic disease progression in the CNS for ≥28 days after definitive radiotherapy and/or surgery.
   * The use of corticosteroids at higher dose occurring ≥28 days prior to the Screening visit unless it is intermittent use for other medical conditions and allowed as a concomitant therapy.
3. Participants with a history of leptomeningeal metastasis are excluded.
4. Prior treatment with an anti-PD-L1 agent (where indicated per protocol) within 5 half-lives.
5. Previous receipt of an Monomethyl auristatin E (MMAE)-containing agent or prior docetaxel.

There are additional inclusion and exclusion criteria. The study center will determine if criteria for participations are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2028-03-10 (Estimated); Study Completion 2032-03-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Approximately 5 years
  Overall survival defined as the time from the date of randomization to the date of death due to any cause.
Progression Free Survival (PFS) assessed by blinded independent central review (BICR) | Approximately 5 years
  Progression-free survival is defined as the time from the date of randomization to the date of the first documentation of objective PD assessed by BICR per RECIST v1.1, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate as assessed by BICR | Approximately 5 years
  The proportion of participants who have a confirmed CR or PR, as best overall response assessed by BICR as per RECIST 1.1.
Progression Free Survival as assessed by Investigator | Approximately 5 years
  Progression Free Survival (PFS) is defined as the time from the date of randomization to the date of the first documentation of objective PD assessed by investigator per RECIST v1.1, or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) as assessed by Investigator | Approximately 5 years
  The proportion of participants who have a confirmed CR or PR, as best overall response assessed by investigator as per RECIST 1.1.
Duration of Response as assessed by BICR | Approximately 5 years
  The time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of the first documentation of PD as determined by BICR assessment per RECIST v1.1, or death due to any cause, whichever occurs first.
Duration of Response as assessed by Investigator | Approximately 5 years
  The time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of the first documentation of PD as determined by investigator assessment per RECIST v1.1, or death due to any cause, whichever occurs first.
Incidence of Treatment Emergent Adverse Events (TEAEs) estimated during the Adverse Events (AE) evaluation | Through 90 days after the last study intervention; Approximately 5 years
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Mean scores and Change from baseline in the global health status/quality of life (QoL) score on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Approximately 5 years
  The EORTC QLQ-C30 is a questionnaire for quantitative measure of health-related quality of life pertinent to participants with a broad range of cancers who are participating in international clinical trials.
Mean scores and Change from baseline in physical functioning and role functioning scores on the EORTC QLQ-C30 | Approximately 5 years
  The EORTC QLQ-C30 is a questionnaire for quantitative measure of health-related quality of life pertinent to participants with a broad range of cancers who are participating in international clinical trials.
Mean scores and Change from Baseline in dyspnea, cough, and chest pain scores on the EORTC Quality of Life Cancer Questionnaire - Lung Cancer 13 QLQ-LC13 | Approximately 5 years
  The EORTC QLQ-LC13 is a lung cancer specific module and consists of 13 item questionnaire assessing lung cancer-associated symptoms and treatment-related effects.
Time to definitive deterioration (TTdD) in in the global health status/QoL score on the EORTC QLQ-C30 | Approximately 5 years
  TTdD is defined as the time from date of randomization to first onset of Patient Reported Outcome (PRO) deterioration without subsequent recovery.
TTdD in physical functioning and role functioning scores on the EORTC QLQ-C30 | Approximately 5 years
  TTdD is defined as the time from date of randomization to first onset of Patient Reported Outcome (PRO) deterioration without subsequent recovery.
TTdD in the dyspnea, cough, and chest pain scores on the EORTC QLQ-LC13 | Approximately 5 years
  TTdD is defined as the time from date of randomization to first onset of Patient Reported Outcome (PRO) deterioration without subsequent recovery.
Pharmacokinetics (PK): Plasma concentration of PF-08046054 and and its components | Approximately 48 weeks
  To characterize the pharmacokinetics (PK) of PF-08046054
Incidence of Anti-Drug Antibody (ADA) | Approximately 48 weeks
  To characterize the immunogenicity of PF-08046054

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (84):
- United States (34):
  - Alabama Oncology, Alabaster, Alabama
  - Alabama Oncology, Bessemer, Alabama
  - Alabama Oncology-, Birmingham, Alabama
  - Alabama Oncology, Birmingham, Alabama
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Cancer Care Centers of Brevard, Inc., Palm Bay, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Illinois Cancer Specialists, Chicago, Illinois
  - Allina Health Cancer Institute - Mercy Hospital, Coon Rapids, Minnesota
  - Allina Health Cancer Institute - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Allina Health Cancer Institute - United Hospital, Saint Paul, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana, Billings, Montana
  - CHRISTUS St. Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Christus St. Vincent Regional Medical Center, Santa Fe, New Mexico
  - White Plains Hospital, White Plains, New York
  - Oncology Hematology Care, Cincinnati, Ohio
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Texas Oncology - Central/South Texas, Austin, Texas
  - Texas Oncology- Central South., Austin, Texas
  - Texas Oncology Central South, Austin, Texas
  - Texas Oncology - Central South (Renfert Way), Austin, Texas
  - Texas Oncology - Dallas (Sammons), Dallas, Texas
  - Texas Oncology- Central South, Harlingen, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - Texas Oncology, McAllen, Texas
  - Texas Oncology- Central South, Waco, Texas
  - Texas Oncology-Central South, Waco, Texas
  - Texas Oncology - Gulf Coast, Webster, Texas
  - Texas Oncology - Central South, Weslaco, Texas
  - Blue Ridge Cancer Care, Blacksburg, Virginia
  - Oncology & Hematology Associates of Southwest Virginia Inc dba Blue Ridge Cancer Care, Salem, Virginia
  - Shenandoah Oncology, P.C., Winchester, Virginia
- Calvary Mater Newcastle, Waratah, New South Wales, Australia
- McGill University Health Centre, Montreal, Quebec, Canada
- China (15):
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jinan Central Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Israel (4):
  - Rabin Medical Center, Petah Tikva, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Sourasky Medical Center, Tel Aviv, TELL ABĪB
- Japan (14):
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure, Hiroshima
  - Hyogo Cancer Center, Akashi, Hyōgo
  - National Hospital Organization Kochi National Hospital, Kochi, Kochi
  - Mie Chuo Medical Center, Tsu, Mie-ken
  - Sendai Kousei Hospital, Sendai, Miyagi
  - National Hospital Organization Nagasaki Medical Center, Ōmura, Nagasaki
  - National Hospital Organization Beppu Medical Center, Beppu-shi, Oita Prefecture
  - NHO Kinki Chuo Chest Medical Center, Sakai, Osaka
  - The University of Osaka Hospital, Suita, Osaka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - National Hospital Organization Tokyo National Hospital, Kiyose, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - National Hospital Organization Okayama Medical Center, Okayama
- Instytut MSF Sp zoo, Lodz, Łódź Voivodeship, Poland
- Ad-Vance Medical Research, Ponce, Puerto Rico
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk-do [chungbuk]
  - Inje University Haeundae Paik Hospital, Haeundae-gu, Pusan-kwangyǒkshi
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
- Hospital Universitario Virgen de Valme, Seville, Spain
- Taiwan (6):
  - Changhua Christian Hospital, Changhua County, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5851005